CLINICAL TRIAL: NCT07071740
Title: Robotic Minimally Invasive Ventral Hernia Repair With DEXTER
Acronym: RAVEN
Status: Completed | Type: Observational
Sponsor: Distalmotion SA (Industry)
Collaborators: Confinis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025-02
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ventral Hernia Repair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ventral hernia repair — Robotic-assisted incisional or primary ventral hernia repair with the DEXTER robotic surgery system

SUMMARY:
The aim of this clinical investigation is to confirm the perioperative and early postoperative safety and clinical performance (efficacy) of the Dexter Robotic System, in patients undergoing incisional or primary ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Planned to undergo incisional and primary midline ventral (M2-M4; epigastric, umbilical and infraumbilical) hernia repair smaller and equal to 8cm
* Patient agrees to perform the 30-day follow-up assessment, as per standard of care

Exclusion Criteria:

* Any planned concomitant procedures
* Active anticoagulant treatment
* Recurring hernia with mesh during primary hernia repair
* Need for transversal abdominal release
* Patients under corticosteroids or other immunosuppressive treatment
* Loss of domain type of hernia
* Previous incision extending from xiphoid process to pubic bone (= Median laparotomy M1 to M5)
* M2 hernia extending to M1 and/or M4 hernia extending to M5
* Ongoing intra-abdominal infection or septic state
* Abdominal fistulae
* History of major* abdominal or pelvic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing incisional or primary ventral hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Primary safety 0utcome | up to 30 days after surgery
  Occurrence of Clavien-Dindo grades III-V adverse events
Primary efficacy outcome | Intraoperative
  Successful completion of the DEXTER-assisted procedure, i.e. free of any conversion to an open or fully laparoscopic surgical approach

CONTACTS AND LOCATIONS:
Locations (5):
- Allgemein öffentliches Krankenhaus Spittal/Drau, Spittal an der Drau, Austria
- GH Saintes - Saint-Jean-d'Angély Site de Saintes, Saintes, France
- Artemed Klinikum München Süd, München, Germany
- Switzerland (2):
  - Kantonsspital Winterthur, Winterthur
  - Hirslanden Klinik Zürich, Zurich